CLINICAL TRIAL: NCT06752876
Title: A Phase 1, Multicenter, Open-Label Study of CB-010, a CRISPR-Edited Allogeneic Anti-CD19 CAR-T Cell Therapy, in Patients With Refractory Systemic Lupus Erythematosus (GALLOP)
Brief Title: CRISPR-Edited Allogeneic Anti-CD19 CAR-T Cell Therapy, in Patients With Refractory Systemic Lupus Erythematosus (GALLOP)
Acronym: GALLOP
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor Strategic Pipeline Prioritization with Focus on CB-010 and CB-011 Oncology Programs
Sponsor: Caribou Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CB10LUPA
Record Dates: First submitted 2024-12-18; First posted 2024-12-31 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Systemic Lupus Erythematosus; Lupus; Lupus Erythematosus; Lupus Nephritis
Keywords: CB-010; Lupus nephritis; Lupus; Extrarenal lupus; Autoimmune disease; Anti-CD19 CAR-T therapy; Cell therapy
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Lupus Nephritis; Autoimmune Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort 1 Lupus Nephritis (LN) (Experimental)
  Interventions: Drug: CB-010
- Cohort 2 Extrarenal Lupus (ERL) (Experimental)
  Interventions: Drug: CB-010

INTERVENTIONS:
Drug: CB-010 — CB-010 allogeneic CAR-T cell therapy, Cyclophosphamide and Fludarabine chemotherapy for lymphodepletion

SUMMARY:
This is a Phase 1 study to evaluate the safety and efficacy of a single infusion of CB-010 in patients with refractory Systemic Lupus Erythematosus (SLE) with cohorts for lupus nephritis (LN) and extrarenal lupus (ERL).

DETAILED DESCRIPTION:
Participants enrolled can expect to be on the study for a total duration of approximately 2 years, during which there will be a screening period followed by a single administration of CB-010 and then 24 months of safety follow-up and monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of SLE according to 2019 EULAR/ACR classification criteria for at least 6 months
* Cohort 1 LN:

  1. Class III or IV lupus nephritis
  2. Urine protein-to-creatinine ratio (UPCR) ≥ 0.8 mg/mg
  3. Refractory to glucocorticoids and at least 2 immunosuppressive therapies
* Cohort 2 ERL (Patients with class I and II LN may be included in the ERL cohort if their SLEDAI-2K is ≥ 8):

  1. SLEDAI-2K ≥ 8
  2. Refractory to glucocorticoids, and at least 2 immunosuppressive therapies
* Adequate renal, hepatic, pulmonary, and cardiac function, with specific laboratory criteria
* Females must be either of nonchildbearing potential, defined as postmenopausal or surgically sterile or agree to use a highly effective double barrier method of contraception or vasectomized partner

Exclusion Criteria:

* Has active severe central nervous system (CNS) lupus in the previous 3 months from planned LD start date
* Has received any other investigational treatment for any indication within the 4 weeks or 5 half-lives
* Prior treatment with cellular therapy (genetically modified cells), gene therapy directed at any target, allogenic or autologous stem cell transplant or organ transplant
* History of infection with human immunodeficiency virus or evidence of hepatitis B or C virus infection
* History of hypersensitivity to Cyclophosphamide, Fludarabine, or any of the components of CB-010
* Received a live vaccine ≤ 6 weeks prior to start of LD
* Patients for whom magnetic resonance imaging (MRI) studies are contraindicated or who cannot tolerate them

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2027-12 (Estimated); Primary Completion 2029-04 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Incidence of critical safety events (CSEs) ≤ 28days after CB-010 infusion | Through 28 days
Incidence of treatment emergent adverse events (TEAEs), serious adverse events (SAEs), and adverse events of special interest (AESIs) | Through end of study (approximately 2 years)

SECONDARY OUTCOMES:
To characterize the PK profile of a single infusion of CB-010 (i.e., CB-010 expansion and persistence) | Through end of study (approximately 2 years)
  Concentration of CB-010 in blood samples over time